CLINICAL TRIAL: NCT03664076
Title: Comiss Score Fore Detection of Cow's Milk Protein Allergy
Brief Title: COMISS Score for Detection of Cow's Milk Protein Allergy in Children With Recrrent or Persistent Gastrointestinal Manifistations in Infants Attending Assuit University Children Hospital - Egypt
Acronym: comiss
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: caroline maher (Other)
Responsible Party: Sponsor-Investigator, caroline maher, internal resident, Assiut University
Organization: Assiut University (Other)
Other Study IDs: AssiutU comiss
Record Dates: First submitted 2018-09-07; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Cow Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: COMISS score — cow's milk protein symptoms score awareness tool to select cow's milk protein allergy in infants

SUMMARY:
COMISS score for detection of Cow's Milk Protein Allergy in children with recurrent or persistent gastrointestinal manifistations in infants attending Assuit University Children Hospital

DETAILED DESCRIPTION:
Cow's-milk protein (CMP) is the leading cause of food allergy in infants and young children younger than 3 years (Sicherer SH.2011) (Rona RJ, et al. 2007).According to a recent meta-analysis, the self-reported lifetime prevalence of cow's milk protein allergy (CMPA)is 6% (range: 5.7-6.4) and the rate of CMPA prevalence defined by the food challenge was 0.6% (0.5-0.8) (Nwaru BI, etal. 2014).Earlier reports estimated an incidence of 2-3% in the first year of life (Høst A. 2002).

CMPA can induce a diverse range of symptoms of variable intensity in infants . Immediate reactions (early) occur from minutes up to 2 hours after allergen ingestion and are more likely to be IgE mediated, whereas delayed reactions (late) manifest up to 48 hours or even 1 week following ingestion. The latter may also involve non-IgE-mediated immune mechanisms. Combinations of immediate and delayed reactions to the same allergen may occur in the same patient.(Shek LP, et al. 2005).

Symptoms and signs related to CMPA may involve many different organ systems mostly the skin and the gastrointestinal and respiratory tracts. The involvement of two systems or more increases the probability of CMPA. Some symptoms are more likely to be present in children with a positive test for CMP-specific IgE (eg. Angioedema and atopic eczema); however, there is a large overlap. The same symptoms may appear in CMP IgE-positive and IgE-negative patients particularly in children with gastrointestinal manifestations (eg, allergic proctitis or proctocolitis) (Shek LP, et al. 2005).

Due to the lack of other reliable diagnostic tests other than a food challenge with CM protein in infants suspected of suffering from cow's milk protein allergy (CMPA), an awareness tool has been developed to recognize cow's milk related symptoms in infants and young children for use by primary healthcare providers. It may help in increasing the awareness and the recognition of cow's milk related symptoms. This tool will help in making decisions and correct management. It would be appreciated by the parents because it will avoid both over and under-diagnosis and also shorten the duration of distress of the infants and parental anxiety. Delayed diagnosis of CMPA has a negative impact on the physical development of children (Robbins KA,et al. 2014) (Vieira MC, et al. 2010) A Cow's Milk-related-Symptom-Score (CoMiSS) is a score that considers general manifestations, dermatological gastrointestinal and respiratory symptoms. It was developed to be used as an awareness tool for cow's milk related symptoms . It can also be used to evaluate and quantify the evolution of symptoms during therapeutic interventions (Vandenplas Y, et al.2015) The CoMiSS score has been shown to be reliable tool in increasing awareness of primary health care physicians to more accurately suspect cow's-milk-related-symptoms.. The findings do suggest that a CoMiSS of >12 may be a good cut-off value to select infants presenting symptoms related to cow's milk protein. The results of the pooled analysis confirm that the CoMiSS may be a sensitive and specific awareness tool for health care professionals to select infants suspected to present with cow's milk related symptoms. A validation trail is still needed to use the score as a diagnostic tool. (YvanVandenplas,et al.2017)

ELIGIBILITY:
Inclusion Criteria:

* Infants of both sex. Age :less than one year attending Assiut university children hospital Persistent ( more than 15 days ) and recurrent ( according to ROM IV criteria ) gastrointestinal manifestations (vomiting, diarrhea, constipation, regurgitation or failure to thrive).

Type of infant feeding: pure breast fed, artificially fed or mixed.

Exclusion Criteria:

* Children older than one year. Infants with acute gastrointestinal manifestations. Previously diagnosed to have any gastrointestinal or systemic disease

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: - Infants of both sex. Age :less than one year attending Assiut university children hospital Persistent ( more than 15 days ) and recurrent ( according to ROM IV criteria ) gastrointestinal manifestations (vomiting, diarrhea, constipation, regurgitation or failure to thrive).
  Type of infant feeding: pure breast fed, artificially fed or mixed
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
COMISS score | one year
  cow's milk protein symptos score

IPD SHARING:
Plan to Share IPD: Undecided